CLINICAL TRIAL: NCT00000743
Title: A Phase I, Dose-Escalating Safety and Tolerance Study of sCD4-PE40 in HIV-Infected Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Upjohn (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 201; 11177 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Alvircept sudotox
Drug: Zidovudine

SUMMARY:
To determine the safety and tolerance of alvircept sudotox (sCD4-PE40) given at various dosing intervals and concentrations. To determine whether frequent dosing alters immunogenicity or toxicity. To obtain preliminary data to ascertain whether sCD4-PE40 has activity against HIV in human subjects. To determine whether there is any additive toxicity with combined use of sCD4-PE40 and zidovudine (AZT).

There is some evidence that AZT and sCD4-PE40, an experimental drug with anti-HIV activity previously demonstrated in vitro, may produce increased benefit when used in combination in HIV-infected patients.

DETAILED DESCRIPTION:
There is some evidence that AZT and sCD4-PE40, an experimental drug with anti-HIV activity previously demonstrated in vitro, may produce increased benefit when used in combination in HIV-infected patients.

Cohorts of six patients each receive escalating doses of sCD4-PE40 in a single IV weekly dose for 8 weeks. All six patients at a given dose must complete 2 weeks of therapy without dose-limiting toxicity before dose escalation in subsequent patient cohorts may occur. The MTD is defined as the dose of sCD4-PE40 immediately below that at which two or more of six patients experience grade 3 or higher toxicity or one or more of six patients experience grade 4 toxicity. After the MTD for the once-weekly schedule is reached, subsequent cohorts receive escalated doses of sCD4-PE40 on a 5x weekly schedule for approximately 4 weeks, in an attempt to establish the MTD for that schedule. When an MTD has been determined for the 5x weekly schedule, and if antiretroviral activity is observed, six additional patients receive this dose combined with AZT for 4 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis with aerosolized pentamidine, trimethoprim / sulfamethoxazole, or dapsone.
* Clotrimazole troches or nystatin oral suspension for oral candidiasis.
* Acyclovir (up to 1000 mg/day for 10 days) for herpes lesions.
* Erythropoietin.

Patients must have:

* Documented HIV infection by ELISA confirmed by a second method. If a prior diagnosis of AIDS has not been established by CDC criteria, a confirmatory test is required.
* CD4 count = or < 300 cells/mm3 within 4 weeks prior to study entry.
* Positive p24 antigen.

Patients entering the AZT portion of the study only:

* Must be AZT naive or have had less than 2 months of AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Hemophilia.
* Acute medical problems (including active opportunistic infections such as active cryptococcosis, Pneumocystis carinii, herpes zoster, histoplasmosis, or CMV or nonopportunistic diseases including liver disease, renal disease, or orthostatic hypotension) at time of study entry.
* Active pulmonary disease.
* Chronic active hepatitis B surface antigenemia or unstable hepatitis C.
* Current diagnosis of malignancy for which systemic therapy would be required during the study.
* Inadequate intravenous access.

Concurrent Medication:

Excluded:

* Hepatotoxic agents.
* Other antiretroviral or immunomodulator agents (including but not limited to AZT, ddI, ddC, interferon, and steroids).
* Other investigational drugs.
* Systemic therapy for malignancy.
* G-CSF and GM-CSF.

Prior Medication:

Excluded:

* Other antiretroviral or immunomodulator agents (including but not limited to AZT, ddI, ddC, interferon, and steroids) within 4 weeks prior to study entry.
* Ribavirin within 90 days prior to study entry.
* Cytotoxic chemotherapy within one month prior to study entry.
* Prior soluble CD4 or CD4-Ig.

Excluded in patients entering the AZT portion of the study:

* More than 2 months of prior AZT therapy.

Current active alcoholism or active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Study Completion 1995-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: van der Horst C, Study Chair
Locations (4):
- United States (4):
  - UCLA CARE Center CRS, Los Angeles, California
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Unc Aids Crs, Chapel Hill, North Carolina

REFERENCES:
- [Background] Alston B, Mitsuyasu R, Lertora J, Flexner C, Timpone J, van der Horst C. Phase I study of sCd4-PE40 in HIV infected persons: (ACTG 201). Int Conf AIDS. 1993 Jun 6-11;9(1):498 (abstract no PO-B29-2178)
- [Background] Fiscus S, et al. Safety and efficacy of soluble CD4-pseudomonas exotoxin 40 in HIV infected individuals (ACTG 201). Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:70